CLINICAL TRIAL: NCT06010342
Title: A Phase 2 Study of TL118 for the Treatment of Patients With Solid Tumors Harboring NTRK Gene Fusions
Brief Title: A Study to Evaluate the Efficacy and Safety of TL118 in Solid Tumors Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Teligene US (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TL-TRK-202101
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor
Keywords: Oncology; TL118; Teligene; Cancer
MeSH Terms: conditions — Neoplasms | interventions — TL-118

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm, Open label (Experimental): Participants will receive TL118 capsule taken orally with (preferred) or without food, 252 mg twice daily, 28 days for a cycle.
  Interventions: Drug: TL118 Capsule

INTERVENTIONS:
Drug: TL118 Capsule — Oral administration

SUMMARY:
The main objective of the study will be to evaluate the efficacy of TL118 in participants with solid tumors harboring NTRK gene fusions

DETAILED DESCRIPTION:
TL118 is an orally active inhibitor of the tropomyosin receptor kinase (Trk) family consists of TrkA, TrkB, and TrkC. These receptors are encoded by the NTRK1, NTRK2 and NTRK3 genes, and oncogenic fusions of NTRK may cause cancer cells to grow and spread in the body. The purpose of this study is to explore how effective TL118 is for the treatment of patients with solid tumors harboring NTRK gene fusions.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years old and above, male or female
2. Histologically or cytologically confirmed diagnosis of locally advanced or metastatic solid tumor that harbors an NTRK1/2/3 gene fusion that is predicted to translate into a fusion protein with a functional tropomyosin receptor kinase (TRK)A/B/C kinase domain, without a concomitant second onco-driver
3. Patients must have had disease progression during or after prior treatment for their tumor, or would be unlikely to tolerate or derive clinical benefit from appropriate standard of care therapy or are not suitable - in the opinion of the Investigator - to receive standard of care therapy; prior treatment with approved or investigational TRK inhibitors is not allowed, except for prior TRK treatment for less than 28 days due to intolerable toxicity)
4. At least one measurable lesion
5. Eastern Cooperative Oncology Group (ECOG) score of 0, 1, or 2
6. A minimum life expectancy of > 3 months
7. Adequate bone marrow reserve, hepatic, renal, and coagulation function

Other inclusion criteria apply for participating in the Study

Exclusion Criteria:

1. Any systemic anti-tumor therapy such as chemotherapy and radiation therapy (including curative radiotherapy or spinal radiotherapy portion > 30%) used within 3 weeks prior to enrollment; immunotherapy within 4 weeks; any palliative radiotherapy for non-target lesions used to relieve symptoms and traditional Chinese medicines (TCMs) indicated for the tumor (including Chinese patent medicine) within 2 weeks prior to enrollment
2. Participation in another interventional clinical trial 2 weeks prior to enrollment or within 5 half-lives from the last dose of IP (whichever is shorter)
3. Any unresolved toxicities from prior therapy greater than Grade 1, at the time of screening with the exception of toxicities posing no safety risk in the opinion of the Investigator
4. Active central nervous system metastases
5. Any other primary malignant tumors within 3 years (except for cured skin basal cell carcinoma and carcinoma in situ of cervix, low-risk cancer
6. Any active infection which has not been controlled at screening

Other exclusion criteria apply for participating in the Study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Pre-dose up to approximately 24 months post-dose

SECONDARY OUTCOMES:
Duration of Response (DoR) | Pre-dose up to approximately 24 months post-dose
Disease Control Rate (DCR) | Pre-dose up to approximately 24 months post-dose
Progression Free Survival (PFS) | Pre-dose up to approximately 24 months post-dose
Time to Tumor Progression (TTP) | Pre-dose up to approximately 24 months post-dose
Time to Response (TTR) | Pre-dose up to approximately 24 months post-dose
Time to Treatment Failure (TTF) | Pre-dose up to approximately 24 months post-dose
Overall Survival (OS) | Pre-dose up to approximately 24 months post-dose
1-year Progression Free Survival | Pre-dose up to approximately 24 months post-dose
1-year Survival | Pre-dose up to approximately 24 months post-dose
Number of Participants Experiencing Adverse Events (AE) | Pre-dose up to approximately 24 months post-dose
Number of Participants Experiencing Adverse Drug Reactions (ADR) | Pre-dose up to approximately 24 months post-dose
Number of Participants Experiencing Serious Adverse Events (SAE) | Pre-dose up to approximately 24 months post-dose
Number of Participants Experiencing Serious Adverse Reactions (SAR) | Pre-dose up to approximately 24 months post-dose
Area Under The Curve (AUC) of TL118 | Pre-dose up to 12 hours post-dose
Maximum Plasma Concentration (Cmax) of TL118 | Pre-dose up to 12 hours post-dose
Minimum Plasma Concentration (Cmin) of TL118 | Pre-dose up to 12 hours post-dose
Time to Peak Drug Concentration (Tmax) of TL118 | Pre-dose up to 12 hours post-dose
TL118 half-life (T1/2) | Pre-dose up to 12 hours post-dose
Apparent Clearance (CL/f) of TL118 | Pre-dose up to 12 hours post-dose
Volume of Distribution (Vz/F) of TL118 | Pre-dose up to 12 hours post-dose

CONTACTS AND LOCATIONS:
Locations (19):
- United States (3):
  - Adventist Health Glendale, Glendale, California
  - Texas Oncology, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- China (16):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University School and Hospital of Stomatology, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou, Guangdong
  - Harbin medical university cancer hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Shanxi Cancer Hospital, Xi'an, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No